CLINICAL TRIAL: NCT04968288
Title: Natural History Study of KSHV-Associated Multicentric Castleman's Disease
Brief Title: Natural History of KSHV-Associated Multicentric Castleman s Disease
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000337; 000337-C
Record Dates: First submitted 2021-07-17; First posted 2021-07-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12-12

CONDITIONS: Multicentric Castleman s Disease
Keywords: Kaposi s sarcoma; HIV; primary effusion lymphoma; interlerleukin-6; Natural History
MeSH Terms: conditions — Lymphoma, Primary Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects with KSHV-associated MCD

SUMMARY:
Background:

Kaposi s sarcoma herpes virus (KSHV) causes several kinds of cancer, Kaposi sarcoma (KS), a form of Multicentric Castleman s Disease (MCD) and a type of lymphoma known as Primary Effusion Lymphoma (PEL). These cancers can occur alone or at the same time in the same patient. MCD can cause a lot of symptoms and problems with various organs in the body, making patients feel quite unwell. If unrecognized, the disease can be fatal. Medications such as rituximab alone or in combination with chemotherapy may help treat MCD but there is little known about the long term effects and the natural course of MCD.

Objective:

To better understand the biology of KSHV-MCD to help identify how this disease causes illness and how cancer treatments known to be effective in MCD may help patients with this condition. This study also aims to help identify ways to treat the disease by providing other standard cancer treatments that would be useful to use to treat MCD based on what we know about this condition.

Eligibility:

People 18 years of age and older with KSHV-MCD.

Design:

Participants will be screened with:

Medical history

Physical exam

CT scan

Blood and heart tests

Participants will have an initial evaluation. This will include:

Review of participants symptoms and ability to perform their normal activities

Blood and urine tests

Imaging studies such as CT and PET scans. Participants may have a contrast agent injected into their arm.

Photographs to document skin lesions

Optional skin biopsy. For this, a small piece of the skin will be removed.

Optional lymph node needle biopsy

Optional samples of the fluid in the space around the lungs, intestines, or heart

Optional sample of the liquid that surrounds the brain and spinal cord

Saliva samples

DEXA scan to examine the bones

Questionnaires

Optional limb measurements or cognitive tests

Physicians will give participants recommendations about treatment.

After their initial evaluation and any treatment, participants will have additional visits. These will occur every 3 months for the first year, then every 6 months for the second year, and then once a year for up to 1 year.

DETAILED DESCRIPTION:
Background:

* Multicentric Castleman s disease (MCD) is a rare but lethal Kaposi s sarcoma-associated herpesvirus (KSHV) associated lymphoproliferative disorder with a historical median survival of 2 years. It occurs more often in HIV-infected individuals than those without HIV infection. The poor prognosis is not fully explained by the underlying HIV, as the HIV-negative cases appear to have little or no survival advantage over the HIV-positive cohort. The disease has no defined standard treatment and there is much to be learned about its pathogenesis and natural history with current treatments.
* Patients with KSHV-MCD may present with other KSHV-associated conditions such as Kaposi sarcoma (KS) and may develop primary effusion lymphoma (PEL) following their diagnosis, which may affect morbidity and mortality. It is not clear how these concurrent conditions develop simultaneously and over time.
* Since 2004, the HIV and AIDS Malignancy Branch (HAMB) has studied the natural history and assessed novel therapies for KSHV-MCD which has contributed to the development of at least two therapies that are now considered as first-line therapies: (1) rituximab plus liposomal doxorubicin and (2) high dose zidovudine plus valganciclovir.
* These therapies plus either rituximab alone or other rituximab-based therapies that have been developed over the last 15 years have resulted in durable responses in patients with KSHV-MCD and have substantially improved the prognosis of these patients.
* The longitudinal evaluations along with tissue sample collection, imaging studies, and participant reported outcomes will allow for the development of a better understanding of the natural history of this disease, and the development of the basis for more effective treatments.

Objective:

-To study and describe the natural history of KSHV-MCD

Eligibility:

* Age >= 18 years
* Biopsy proven KSHV-associated MCD

Design:

* This will be a long-term study to comprehensively study participants with KSHV-MCD
* Medical history will be collected, and participants followed throughout the course of their illness, with particular attention to patterns of disease presentation, recurrence and progression, response to therapies, and duration of responses
* Tissue samples and blood will be obtained from participants during this study.
* We anticipate accruing 135 evaluable participants on this protocol

ELIGIBILITY:
* INCLUSION CRITERIA:
* Biopsy proven KSHV-associated MCD, confirmed in the Laboratory of Pathology (LP), CCR
* Age >=18 years.
* ECOG performance status <=4 (Karnofsky >=20%).
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Participants may be co-enrolled in other protocols, including investigational studies to treat KSHV-associated malignancies.

EXCLUSION CRITERIA:

* Any condition or set of circumstances that in the opinion of the investigators would make participation in this study unsafe or otherwise inappropriate for a given individual.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2034-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
natural history of MCD | ongoing
  clinical presentation, patterns of disease progression, therapeutic response, disease recurrence and participant overall survival

SECONDARY OUTCOMES:
concurrent KS or PEL evaluation | every 3 months for year 1, every 6 month for year 2, yearly from year 3
  Percentage of subjects with concurrent PEL or KS
relapse-free survival | every 3 months for year 1, every 6 month for year 2, yearly from year 3
  time from any treatment until first recurrence
overall survival | every 3 months for year 1, every 6 month for year 2, yearly from year 3
  time from any treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Ramya M Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000337-C.html